CLINICAL TRIAL: NCT03294109
Title: Evaluation of Abdominal Wall Block With Liposomal Bupivacaine for Post-Operative Analgesia in Donor Nephrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Siamak Rahman, MD, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-000598
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Pain, Postoperative; Analgesics, Opioid; Analgesics, Non-Narcotic; Physiological Effects of Drugs; Peripheral Nervous System Agents; Patient Satisfaction; Return to Work; Activity, Sexual
Keywords: TQL block, TAP block, donor nephrectomy, pain, patient satisfaction
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Sexual Behavior; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- study (Experimental): liposomal bupivacain
  Interventions: Drug: Abdominal wall block with liposomal bupivicaine
- control (No Intervention): no intervention

INTERVENTIONS:
Drug: Abdominal wall block with liposomal bupivicaine — Abdominal wall block with liposomal bupivicaine
  Other Names: Exparel
  Arms: study

SUMMARY:
A blinded randomized control trial in living kidney donors. The study group will receive a liposomal bupivacaine Trans Quadratus Lumborum (TQL) block after the induction of general anesthesia. The following study variables will be collected postoperatively following arrival in the post-anesthesia care unit. Current and maximum intensity pain scores will be documented by nurses in Electronic Health Record (EHR). Total opiate dose consumed every 24 hours will be collected from the EHR and pain diary after discharge. Patient satisfaction will be evaluated using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) 24 hours' post-procedure. Incidence of nausea will be extracted from nursing notes.

DETAILED DESCRIPTION:
This is a blinded (patients are blinded and all the staff and the nurses who collect data are also blinded) randomized controlled trial in living kidney donors who have been approved by a multidisciplinary (nephrology, urology, psychiatry, and social work) team to proceed with donor nephrectomy. Patients will be approached to participate in the study only after they have agreed to kidney donation and have been informed of all of the associated risks. Participants are informed that they can withdraw from kidney donation at any time until they are in the operating room.

Patients meeting these criteria, who also consent to participate in the study, will be randomized (standard of care pain medication vs TQL block). The ratio of male to female patients in each arm will be equal because of the known increased risks for post-operative nausea/vomiting (PONV) in females. The study group will receive a liposomal bupivacaine TQL block after the induction of general anesthesia and liposomal bupivacaine transverse abdominis plane (TAP) block after closure of the midline fascia. All patients including the control group will have infiltration of the skin edges with bupivacaine. Control patients will have a TAP block with 5 cc of bupivacaine on both sides. A placebo 22g needle will be placed at the same site as the TQL block without injection. Intra-operative narcotics will be administered by the anesthesia team based on standard criteria. All participants will receive intravenous ketorolac and acetaminophen at the end of the procedure. Intravenous ketorolac will be continued for 24 hours while hospitalized. Post-operative pain management with intermittent parenteral and enteral narcotics as needed will be the same in both groups.

Liposomal bupivacaine block administration:

After induction of general anesthesia, surgical team will turn the patient to the lateral position (final position for surgery). After prep with and drape, investigators will place ultrasound probe in mid- posterior axillary line, just above iliac crest. The investigators will identify abdominal wall muscles including external oblique, internal oblique, transverse abdominis, and quadratus lumborum as well as thoracolumbar fascia with the help of ultrasound. Then, investigators will insert a 22g nerve block needle and advanced it under direct guidance of ultrasound until it is below the fascial covering of the quadratus lumborum muscle layer or its fascia which forms a continuous fascia compartment with thoracolumbar fascia. After aspiration to rule out intravascular location of the needle, investigators will be inject 20 mL of liposomal bupivacaine mixed with 10ml of normal saline under ultrasound guidance, to monitor spread of the injected fluid . The investigators will aspirate repeatedly every 5cc of local anesthetic. The investigators will remove the needle upon completion of the injection.

The following study variables will be collected postoperatively following arrival in the post-anesthesia care unit. Current and maximum intensity pain scores will be documented by nurses in EHR. Total opiate dose consumed every 24 hours will be collected from the EHR and pain diary after discharge. Patient satisfaction will be evaluated using the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) 24 hours' post-procedure. Incidence of nausea will be extracted from nursing notes

Complications will be documented by anesthesia pain service that will follow these patients while admitted.

Outpatient use of narcotics, pain assessment, bowel function, sexual function complications from the block or the donor surgery, and attitudes toward kidney donation will be evaluated with validated survey instruments. Please see the timeline for the collection of the data prior to and after kidney donation. The survey data will be collected using secure links to a REDCap server 3, 5, 10, 30, and 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic donor nephrectomy

Exclusion Criteria:

* Pregnancy
* Systemic or local infection at the potential block site.
* Allergy or hypersensitivity to the local anesthetic,
* Possible variations in surgical approach to donor nephrectomy other than what is defined in this protocol.
* Scarring or anatomic abnormality over the proposed injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Rahman, MD, Principal Investigator — University of California, Los Angeles; Hans a Gritsch, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Connie Frank Kidney Transplant Center, Los Angeles, California, United States

REFERENCES:
- [Background] Wikner M. Unexpected motor weakness following quadratus lumborum block for gynaecological laparoscopy. Anaesthesia. 2017 Feb;72(2):230-232. doi: 10.1111/anae.13754. Epub 2016 Nov 28. PMID 27891579
- [Background] Dam M, Moriggl B, Hansen CK, Hoermann R, Bendtsen TF, Borglum J. The Pathway of Injectate Spread With the Transmuscular Quadratus Lumborum Block: A Cadaver Study. Anesth Analg. 2017 Jul;125(1):303-312. doi: 10.1213/ANE.0000000000001922. PMID 28277325
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Background] Hansen CK, Dam M, Bendtsen TF, Borglum J. Ultrasound-Guided Quadratus Lumborum Blocks: Definition of the Clinical Relevant Endpoint of Injection and the Safest Approach. A A Case Rep. 2016 Jan 15;6(2):39. doi: 10.1213/XAA.0000000000000270. No abstract available. PMID 26771297
- [Derived] Gritsch HA, Osbun N, Grogan T, Fero KE, Partownavid P, Stockman J, Sadoughi N, Park E, Miller E, Blumberg J, McDonald M, Cowan N, Shah N, Rahman S. Randomized controlled trial of a quadratus lumborum block with liposomal bupivacaine for postoperative analgesia in laparoscopic donor nephrectomy. Clin Transplant. 2021 Sep;35(9):e14403. doi: 10.1111/ctr.14403. Epub 2021 Jul 14. PMID 34184312
- See also: Quadratus lumborum block: an effective method of perioperative analgesia in children undergoing pyeloplasty — http://dx.doi.org/10.1016/j.jclinane.2015.05.006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, 146 patients signed consent. Of those 146, 137 completed the intake questionnaire, a requirement for the study. Of those 137, 103 were scheduled for surgery.
Groups:
- Study: ERAS Plus laparoscopic TAP block and transmuscular quadratus lumbarum with liposomal bupivicaine:
- Control: ERAS Plus laparoscopic TAP block
Period: Overall Study
Arm/Group | Study | Control
Started | 46 | 57
Underwent Surgery | 40 | 52
Completed | 40 | 52
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Study: ERAS Plus laparoscopic TAP block and transmuscular quadratus lumbarum with liposomal bupivicaine
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 40 | 52 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 49 | 86
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 64
  Male | 12 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 27 | 33 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 13 | 18
Region of Enrollment [Number; unit: participants]
  United States | 40 | 52 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Visual Analog Score (VAS) for pain, scores range from 0-10, with lower scores indicating lower pain level
Time Frame: 3 days post-op
Population: Participants who completed pain VAS survey on day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 25 | 36
score on a scale | 4.20 (1.94) | 4.62 (1.74)

2. Secondary Outcome: Patient Satisfaction With Pain Management
Description: The Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) survey score on variable "Satisfaction with Pain Treatments." This is a scale ranging from 0-10, with 0 being extremely dissatisfied, a poor outcome, with pain treatment to 10 being extremely satisfied, a better outcome.
Time Frame: Day 1
Population: Patients who completed APS-POQ-R survey question "Satisfaction with Pain Treatments" on Day 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 39 | 46
score on a scale | 8.6 (1.9) | 9.1 (1.2)

3. Secondary Outcome: Nausea and Vomiting, Defined as Requiring Pre-op Scopolamine Patch or Rescue Antiemetics
Description: Number of patients requiring pre-op scopolamine patch, and number of patients requiring rescue antiemetics in PACU.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 40 | 52
Participants
  pre-op Scopolamine patch | 9 | 11
  Rescue antiemetics in PACU | 6 | 8

4. Secondary Outcome: Return of Bowel Function
Description: Bowl activity survey asked participants how big a problem the bowel function was after surgery, on a scale of 1 (no problem) to 5 (a big problem).
Time Frame: Day 5
Population: Participants who completed the bowel activity survey on Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study | Control
Number analyzed (Participants) | 31 | 38
score on a scale | 1.9 (1) | 1.9 (1.1)

5. Secondary Outcome: Participants Experiencing Complications Related to Surgery or Block
Description: Number of participants that experienced a related complication in each arm
Time Frame: Duration of inpatient stay, up to 5 days
Population: All enrolled patients receiving surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 42 | 50
Participants | 5 | 3

6. Secondary Outcome: Opioid Use Dose/Day
Description: Milligram Morphine Equivalent /day
Time Frame: Day 3
Population: Patients whom responded to survey on Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 25 | 29
Participants
  0 MME | 11 | 9
  >0 - 5 MMe | 6 | 8
  >5 - 10 MME | 3 | 8
  >10-15 MME | 3 | 2
  >15-20 MME | 2 | 1
  >20 MME | 0 | 1

ADVERSE EVENTS:
Time Frame: During hospitalization, up to 5 days
Description: Complications from surgery were collected as adverse events.
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/50
Other Adverse Events (participants affected / at risk) | 5/42 | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study (N=42) | Control (N=50)
Urinary Retention (Renal and urinary disorders) | 1 | 1
Pleural Effusion requiring aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Incisional hematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound infection (Injury, poisoning and procedural complications) | 1 | 0
Contralateral flank pain and acute kidney injury (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Blood and lymphatic system disorders) | 1 | 0 — Post-operative hypotension in setting of acute blood loss
Wound seroma (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03294109/Prot_SAP_000.pdf